CLINICAL TRIAL: NCT05655780
Title: Optimal Survival and Quality of Life in Patients With Metastatic Colorectal Cancer With Irinotecan Dosing Based on UGT1A1 Genotype and Gut Microbiota Enzyme Activity Including a Dietary Intervention (OPTIMA)
Brief Title: The Role of the Tumor Molecular Profile (CMS), UGT1A1 Genotype and Beta-glucuronidase Activity of the Intestinal Microbiota for Treatment Efficiency, Toxicity, Survival and Quality of Life in Patients With Metastatic or Unresectable Colorectal Cancer During Irinotecan-based Systemic Treatment
Acronym: OPTIMA
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Maastricht University (Other); Wageningen University & Research (Unknown); Fontys Hogeschool (Unknown); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Erasmus Medical Center (Other); Catharina Ziekenhuis (Unknown); University of North Carolina (USA) (Unknown); Oncology patientenpanel MUMC (Unknown); Stichting Kanker.nl (Unknown); Van Weel-Bethesda Ziekenhuis (Unknown); VieCuri Medisch Centrum voor Noord-Limburg (Unknown); Gelderse Vallei Hospital (Other); Danone Nutricia Research (Industry); Clinical Trial Center Maastricht B.V. (Other); Dutch Colorectal Cancer Group (DCCG) (Unknown); Prospectief Landelijk CRC Cohort (PLCRC) (Unknown); CRC-guideline committee (Unknown); CZ zorgverzekeraar (Unknown); Landelijke Werkgroep Diëtisten Oncologie (LWDO) (Unknown); Rode Kruis Ziekenhuis Beverwijk (Unknown)
Responsible Party: Sponsor
Other Study IDs: METC 2022-3247
Record Dates: First submitted 2022-12-08; First posted 2022-12-19 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Irinotecan-based systemic therapy is a treatment option for metastatic or unresectable colorectal cancer. However, this therapy has two major disadvantages, namely, an unpredictable response to the treatment and severe side effects, for instance diarrhea or a low white blood cell count (neutropenia). Therefore, the OPTIMA study was developed to find out if biomarkers, such as the molecular profile of the tumor, the UGT1A1 genotype and activity of the bacterial enzyme β-glucuronidase, can predict response and side effects during irinotecan treatment. By looking at these biomarkers, treatments could be more personalized, resulting into enhanced therapy efficiency, increased optimal survival and a better quality of life.

DETAILED DESCRIPTION:
Irinotecan-based systemic therapy is shown to have promising results in metastatic or unresectable colorectal cancer. However, this therapy has two major disadvantages, including an unpredictable individual treatment response and late-onset systemic and gastrointestinal toxicity. To target these problems, biomarkers are needed which could be used to predict treatment response and toxicity before start of the treatment. The molecular profile of the tumor (consensus molecular subtypes (CMS)), the UGT1A1 genotype and the gut microbiota-derived enzyme β-glucuronidase are promising candidates in this context. Recent research demonstrated that irinotecan-based systemic therapy increased both progression free survival (PFS) and optimal survival (OS) predominantly in patients with CMS4 cancers, as well as in preclinical models representing this subtype. For the other CMS subtypes (CMS1-3), irinotecan-based systemic therapy was shown to be significantly less efficient. For the UGT1A1 genotypes, decreased activity of the UGT1A1 enzyme (converting the toxic metabolite SN-38 into the inactive SN-38G) will increase the concentration of toxic SN-38, resulting in systemic toxicity. Lastly, the importance of studying bacterial β-glucuronidase (β-GUS) activity in CRC patients during treatment with irinotecan can be derived from recent animal studies, and indirect human evidence. Previous research has shown that high bacterial β-GUS activity (converting the inactive SN-38G into the toxic SN-38) might be a possible indicator for irinotecan-induced late-onset gastrointestinal toxicity due to SN-38 accumulation. Therefore, the OPTIMA study was developed to combine prediction of tumor sensitivity towards irinotecan (by CMS classification), UGT1A1 expression for irinotecan dose determination, and β-GUS for risk assessment for late-onset gastrointestinal toxicity. The aim of the study is to investigate whether the molecular profile of the tumor (e.g. based on CMS), the UGT1A1 genotype and β-GUS activity can act as a predictor for therapy efficiency, late-onset systemic and gastrointestinal toxicity, as well as OS and quality of life (QoL).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient: 18 years of age or older
* Patients diagnosed with metastatic or unresectable CRC, who will be treated with irinotecan-based systemic therapy with or without anti-eGFR treatment.
* WHO performance status 0-2
* Minimal acceptable safety laboratory values defined as:

  * ANC of ≥ 1.5 x 109 /L
  * Platelet count of ≥ 100 x 109 /L
  * Hepatic function as defined by serum bilirubin ≤ 1.5 x ULN, ALAT and ASAT ≤ 2.5 x ULN; in case of liver metastases ALAT and ASAT ≤ 5 x ULN.
  * Renal function (eGFR) ≥ 50 ml/min or OR creatinine ≤ 1.5 x ULN
* Written informed consent

Exclusion Criteria:

* Microsatellite instability (MSI) or deficient MMR proteins
* Pregnant or nursing
* Presence of ileostomy
* Asian ethnicity
* Other systemic treatment is less than one month before the start of the irinotecan-based treatment
* Therapeutic antibiotic use is less than three months before the start of the irinotecan-based treatment
* Abdominal radiotherapy is less than two weeks before the start of the irinotecan-based treatment
* Physically or mentally incapable or incompetent
* More than 25% irinotecan dose reduction at the start of treatment (dose reductions during treatment are allowed), with exception of dose reduction due to UGT1A1 mutation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 104 participants will be included for this study. The patients will be addressed for participation in several hospitals in the Netherlands, including the Maastricht University Medical Centre+, Catharina Hospital, Amsterdam UMC, Hospital Gelderse Vallei, Van Weel-Bethesda Hospital and VieCuri Hospital. All participants are asked to sign an informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Bacterial beta-glucuronidase activity | 2022-2028
  Bacterial beta-glucuronidase activity will be measured in faecal samples by using a validated beta-glucuronidase enzyme activity assay, which is based on previous studies. If we measure beta-glucuronidase activity, we will be able to predict late-onset gastrointestinal toxicity because we can estimate the amount of toxic SN-38 that will be produced.
UGT1A1 (uridine diphosphate glucuronosyltransferase) | 2022-2028
  UGT1A1 will be measured by using blood samples, since decreased activity of the UGT1A1 enzyme will ensure an increase in toxic SN-38. When we measure the activity of the UGT1A1 enzyme, we can adjust the treatment dose based on this and, consequently, reduce gastrointestinal toxicity.
Molecular profile of the tumor | 2022-2028
  Associations between the baseline molecular profile of the tumor (e.g. CMS) and response to irinotecan-based treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marjolein Smidt, Prof. dr., Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht UMC+, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Russ E, Ziemons J, Hillege LE, van Kuijk SMJ, de Jong EM, Elbers C, Deenen MJ, Borghuis LH, Bohm TMM, Kristen P, Valk LC, van Hellemond IEG, Vestjens H, Dietvorst A, Baars A, Goosens ANM, Vermeulen L, Buffart TE, de Vos-Geelen J, Penders J, Redinbo MR, Iersel LV, Smidt ML. Evaluation of potential biomarkers during irinotecan-based systemic treatment for colorectal cancer-study protocol of the OPTIMA study. BMC Cancer. 2025 Jul 1;25(1):1129. doi: 10.1186/s12885-025-14500-6. PMID 40597074